CLINICAL TRIAL: NCT05987228
Title: Effects of Orally Administered Thymus Vulgaris Leaves on Memory, Anxiety, Depression, and Sleep Quality in University Students: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hashemite University (Other)
Responsible Party: Principal Investigator, Abdelrahim Alqudah, Assisstant professor, The Hashemite University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 22/6/2022/2023
Record Dates: First submitted 2023-08-01; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Memory Dysfunction; Anxiety; Depression; Sleep
Keywords: Thymus vulgaris leaves; Memory performance; Anxiety; Depression; Sleep
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thymus vulgaris group (Experimental): 500 mg of Thymus vulgaris (capsules) was given orally twice daily
  Interventions: Dietary Supplement: Thymus vulgaris
- control group (Placebo Comparator): 500 mg starch (capsules) was given orally twice daily
  Interventions: Dietary Supplement: Thymus vulgaris

INTERVENTIONS:
Dietary Supplement: Thymus vulgaris — 500 mg of Thymus vulgaris (capsules) was given orally twice daily

SUMMARY:
Thymus vulgaris could potentially serve as a safer alternative to stimulant drugs for enhancing memory among university students. Furthermore, Thymus vulgaris may offer additional benefits in terms of reducing anxiety, depression, and improving sleep quality. However, it should be noted that the current research on the effects of orally administered Thymus vulgaris on the brain and nervous system is limited, and further studies are required to fully explore its potential advantages. Therefore, the purpose of this study is to investigate the effects of oral Thymus vulgaris on memory performance, anxiety, depression, and sleep quality in university students.

DETAILED DESCRIPTION:
Thymus vulgaris belongs to the Lamiaceae family and is a flowering plant. It can be found worldwide, although its origin is in southern Europe [1]. This plant is characterized by its compact, bushy nature and evergreen shrub structure. Its leaves are small, gray-green, highly aromatic, and it produces clusters of purple or pink flowers [2]. Thymus vulgaris is commonly used as a spice to enhance the flavor of food. It is also utilized in the form of dietary supplements; such as capsules or essential oils [3]. Throughout history, Thymus vulgaris has been employed in folk medicine due to its remarkable antimicrobial and anti-inflammatory properties [4]. In Jordanian traditional medicine, it is frequently utilized as an antiseptic, bronchial, sedative, and spasmolytic agent, as well as to improve cognitive function and memory [5-8]. Numerous studies have reported various health benefits associated with Thymus vulgaris leaves, including antioxidant [9], diuretic [10], anti-inflammatory [11], antiviral [12], anti-cancerous [13], cholesterol-lowering [14], glucose-lowering [15], anticonvulsant [16], anti-anxiety [17] and sedative-hypnotic activities [18].

The primary constituents of Thymus vulgaris, notably thymol, p-cymene, γ-terpinene, linalool, and carvacrol, possess various neuropharmacological properties, including anti-anxiety, sedative, anticonvulsant, memory-enhancing, and anti-Alzheimer's disease effects [19]. Asadbegi et al. conducted a study demonstrating that thymol exhibited neuroprotective properties by reducing memory impairment caused by intrahippocampal injection of the amyloid beta (Aβ) peptide in rats fed a high-fat diet [20]. Furthermore, Capibaride et al. confirmed the significant antidepressant-like effect of thymol by observing its ability to reverse behaviors associated with chronic corticosterone exposure and decrease in BDNF levels in female mice [21]. Azizi et al. demonstrated that carvacrol and thymol exerted neuroprotective effects against Aβ25-35-induced damage, potentially through the attenuation of oxidative stress and the modulation of PKC activity, a protein associated with memory function [22]. Additionally, within the monoterpenes and sesquiterpenes, β-myrcene and caryophyllene have been identified as major compounds. β-myrcene is known for its analgesic, anxiolytic, and anti-inflammatory effects [23].

Multiple studies have highlighted the positive impact of Thymus vulgaris on memory, anxiety, and depression. Akan et al. conducted research on rats using the Morris water maze and found that Thymus vulgaris L. exhibited beneficial effects against diabetes mellitus-induced neuropathy and cognitive impairment [24]. They attributed these effects to specific components like thymol, carvacrol, 8-terpinene, p-cymene, and α-pinene present in high amounts in the essential oil composition. Similarly, Rabiei et al. suggested that Thymus vulgaris extract demonstrated anti-amnesic properties in rats with Sco-induced memory deficits, as assessed by the Morris water maze and passive avoidance tests [25]. The authors proposed that this effect could be linked to the extract's antioxidant activity or its influence on the cholinergic system, with carvacrol and thymol playing significant roles based on their chemical composition. Additionally, an ethanol extract derived from Thymus vulgaris leaves displayed an anxiolytic profile in rats during the EPM test, unaffected by locomotor activity [17]. Finally, in the context of Alzheimer's disease, a neurodegenerative disorder involving cholinergic neuron loss, administration of thyme oil to Caenorhabditis elegans enhanced neurotransmission by regulating synaptic acetylcholine levels [26].

The high prevalence of anxiety, depression, and sleep disorders among university students can significantly affect their memory function [27]. Consequently, an increasing number of university students have turned to using stimulant drugs to improve their memory performance and attention, despite the fact that such usage is unauthorized and not intended for therapeutic purposes [28]. However, the use of these drugs is associated with various side effects[29,30]. This has led neuroscience researchers to show a growing interest in identifying cognitive-enhancing drugs that can be safely used by healthy individuals without any detrimental effects.

Based on the provided information, it is hypothesized that Thymus vulgaris could potentially serve as a safer alternative to stimulant drugs for enhancing memory among university students. Furthermore, Thymus vulgaris may offer additional benefits in terms of reducing anxiety, depression, and improving sleep quality. However, it should be noted that the current research on the effects of orally administered Thymus vulgaris on the brain and nervous system is limited, and further studies are required to fully explore its potential advantages. Therefore, the purpose of this study is to investigate the effects of oral Thymus vulgaris on memory performance, anxiety, depression, and sleep quality in university students.

ELIGIBILITY:
Inclusion Criteria:

* Health participants

Exclusion Criteria:

* individuals with medical diseases, psychiatric disorders, those using any medications (including complementary and alternative medicines), as well as pregnant and lactating individuals, were excluded from participating

Ages: 19 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Memory performance | 30 days
  Prospective and Retrospective Memory Questionnaire (PRMQ) was employed

SECONDARY OUTCOMES:
Anxiety and depression | 30 days
  Anxiety and depression levels were measured using the Hospital Anxiety and Depression Scale (HADS)
Sleep quality | 30 days
  Pittsburgh Sleep Quality Inventory (PSQI) questionnaire was performed

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pharmaceutical Sciences, Zarqa, Jordan